CLINICAL TRIAL: NCT04775290
Title: Monocentric, Randomized Clinical Trial About the Effect of Yoga Practice on QOL, Physiological Distress and Fatigue, on Patients Affected by Breast Cancer Undergoing Adjuvant Radiotherapy
Brief Title: Yoga on QOL Physiological Distress&Fatigue, on Patients Affected by Breast Cancer in Adjuvant Radiotherapy
Acronym: YogaRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRST174.21
Record Dates: First submitted 2020-12-14; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Female Breast Cancer; Fatigue; Quality of Life; Physiological Stress; Radiotherapy; Complications
Keywords: Female Breast Cancer; Fatigue; Quality of Life; Physiological Stress; Radiotherapy; Complications
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Yoga (YG) (Experimental): Patients assigned to the YG arm participate in yoga classes
  Interventions: Behavioral: Yoga lessons
- Arm control (CG) (No Intervention): Patients assigned to the CG arm will follow the normal course of radiotherapy.

INTERVENTIONS:
Behavioral: Yoga lessons — 2 weekly yoga classes during the 5 weeks of radiotherapy
  Arms: Arm Yoga (YG)

SUMMARY:
The study aims to investigate, through serial measurements of some biomarkers, the potential mechanisms through which yoga impacts on QOL and fatigue.

DETAILED DESCRIPTION:
The study aims to assess QoL, fatigue and physiological distress (cortisol and proinflammatory markers) with blood sampling on day 1,15 and last of radiotherapy, at 1-3-6 months after the end of radiotherapy.

Patients with breast cancer who will undergo radiotherapy will be randomly assigned to the yoga group (YG) or the control group (CG).

Patients in the YG will participate in 2 weekly yoga classes during the 5 weeks of radiation therapy. The classes will be coordinated with the treatment program and will be held in the vicinity of the radiation therapy center.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage 0-III breast cancer who have undergone adjuvant daily radiotherapy for 5 weeks in Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori (IRST) Department of Radiation Oncology of Meldola.

Exclusion Criteria:

* Patients with documented diagnosis of mental disorders (eg Schizophrenia)
* Patients with stage IV disease
* Patients with active or non-canalised deep vein thrombosis
* Patients not undergoing surgery for the basic oncological disease
* Patients with mobility problems (eg unable to get up from the chair)
* Patients who have practiced yoga or are practicing yoga in the 6 months before the cancer diagnosis.
* Patients diagnosed with lymphedema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 120 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-04-04 (Estimated)

PRIMARY OUTCOMES:
Change of physiological distress | up to 32 months
  Evaluation of the efficacy of yoga on reduction of physiological distress after the end of radiotherapy, measured via Short Form 36 (SF-36), Pittsburgh Sleep Quality Index (PSQI) and Quality of life questionnaire Core30 (QLQ-C30) questionnaire, and physiological functions (cortisol, blood sampling with proinflammatory markers evaluation) in stage 0-III breast cancer patients

SECONDARY OUTCOMES:
Evaluation of quality of life with yoga during and after radiotherapy | up to 6 months
  Assess whether yoga helps on increase Quality of Life (QOL) and decreasing fatigue via questionnaire Brief Fatigue Inventory (BFI).

CONTACTS AND LOCATIONS:
Overall Officials: Simona Micheletti, MD, Principal Investigator — IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l.
Locations (1):
- IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST s.r.l., Meldola, Forlì-Cesena, Italy

REFERENCES:
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669